CLINICAL TRIAL: NCT01927081
Title: Self-management Interventions for Pain in Advanced Breast Cancer
Brief Title: Self-management Interventions for Advanced Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00044446
Record Dates: First submitted 2013-08-16; First posted 2013-08-22 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Advanced Breast Cancer Stage IV

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- discussion group (Active Comparator): Eight weekly group sessions in which participants will engage in discussions regarding issues related to coping with advanced cancer and pain
  Interventions: Behavioral: discussion group
- discussion group + exercise (Active Comparator): Eight weekly group sessions in which participants will engage in discussions regarding issues related to coping with advanced cancer and pain and learn gentle exercise and breathing techniques
  Interventions: Behavioral: discussion group; Behavioral: gentle exercise

INTERVENTIONS:
Behavioral: discussion group — Participants engage in discussions regarding issues related to coping with advanced cancer and pain
Behavioral: gentle exercise — Patients learn gentle exercise and breathing techniques
  Arms: discussion group + exercise

SUMMARY:
The purpose of this research study is to evaluate whether self-management discussion groups are helpful for women with advanced breast cancer who are experiencing pain. The study is looking at the usefulness of two different types of discussion groups, one of which also includes gentle exercise.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Stage IV breast cancer or recurrent metatastic breast cancer
* receiving care at Duke Cancer Institute,
* life expectancy ≥9 months as estimated by the treating oncologist,
* speak and read English,
* be at least age 18
* be able to travel to the Duke Cancer Institute

Exclusion Criteria:

* cognitive impairment as assessed by the 6-item Mini-mental Status Exam,
* Karnofsky Performance Rating of <60 as rated by the oncology provider, an ECOG rating of 0-2
* treatment for serious psychiatric illness (e.g., schizophrenia, severe depression) in the past 6 months,
* currently engaged in yoga practice ≥ 1 day per week

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2014-09; Primary Completion 2017-11-20 (Actual); Study Completion 2017-11-20 (Actual)

PRIMARY OUTCOMES:
Feasibility | 36 months
  Feasibility will be indicated by our ability to meet accrual goals, and by at least 70% of patients attending ≥4 of 8 sessions and providing post-test assessments
Acceptability | 36 months
  Acceptability will be assessed via participant ratings on a standardized measure of treatment effectiveness/satisfaction, supplemented by exit interview

SECONDARY OUTCOMES:
Change in pain | study entry, following completion of the intervention (approximately 3 months), 6 months, and 9 months
  pain intensity as assessed by the Brief Pain Inventory
Change in fatigue | study entry, following completion of the intervention (approximately 3 months), 6 months, and 9 months
  Fatigue as assessed by the Brief Fatigue Inventory
Change in sleep disturbance | study entry, following completion of the intervention (approximately 3 months), 6 months, and 9 months
  Sleep disturbance as assessed by the Pittsburgh Sleep Quality Index
Change in Psychological distress | study entry, following completion of the intervention (approximately 3 months), 6 months, and 9 months
  Anxiety and depression assessed using the Hospital Anxiety and Depression Scale
Change in functional capacity | study entry, following completion of the intervention (approximately 3 months), 6 months, and 9 months
  Functional capacity assessed using a 6-minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Laura Porter, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Carson JW, Carson KM, Olsen MK, Sanders L, Porter LS. Mindful Yoga for women with metastatic breast cancer: design of a randomized controlled trial. BMC Complement Altern Med. 2017 Mar 13;17(1):153. doi: 10.1186/s12906-017-1672-9. PMID 28288595